CLINICAL TRIAL: NCT02792803
Title: An 8 Week Comparison of Xalatan (Latanoprost) to Apo-latanoprost and Co-latanoprost in the Treatment of Open Angle Glaucoma
Brief Title: A Comparison of Xalatan (Latanoprost) to Apo-latanoprost and Co-latanoprost in the Treatment of Glaucoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. David Yan (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Dr. David Yan, M.D., F.R.C.S. (C), DBYAN Medicine Professional Corporation
Organization: DBYAN Medicine Professional Corporation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00012759
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: POAG; Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: POAG; Primary open angle glaucoma; Ocular Hypertension; Xalatan; Latanoprost; Ocular Hyperemia; IOP; Intraocular Pressure; Allergan; prostaglandin
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xalatan --> Apo-/Co-Latanoprost (Experimental): Patients in this arm will be prescribed Xalatan for the first four week period of the study and one of the generics, Apo- or Co-Latanoprost, for the second four week period. Patients will take one drop of the assigned drops in the affected eye every evening at 2100 hrs (+- 1 hr)
  Interventions: Drug: Xalatan; Drug: Apo-Latanoprost; Drug: Co-Latanoprost
- Apo-/Co-Latanoprost --> Xalatan (Experimental): Patients in this arm will be prescribed one of the generics, Apo- or Co-Latanoprost, for the first four week period of the study and Xalatan for the second four week period. Patients will take one drop of the assigned drops in the affected eye every evening at 2100 hrs (+- 1 hr)
  Interventions: Drug: Xalatan; Drug: Apo-Latanoprost; Drug: Co-Latanoprost

INTERVENTIONS:
Drug: Xalatan — A prostaglandin analogue used to reduce intraocular pressure in patients diagnosed with glaucoma.
  Other Names: 02231493; Latanoprost
Drug: Apo-Latanoprost — A prostaglandin analogue used to reduce intraocular pressure in patients diagnosed with glaucoma.
  Other Names: 02296527
Drug: Co-Latanoprost — A prostaglandin analogue used to reduce intraocular pressure in patients diagnosed with glaucoma.
  Other Names: 02254786

SUMMARY:
The purpose of the study is to provide evidence that the efficacy of Xalatan will be superior to Apo-latanoprost and Co-latanoprost in the reduction of intraocular pressure in patients with primary open angle glaucoma. The study will also aim to prove the tolerability of Xalatan in terms of ocular hyperemia will be equivalent to its generic counterparts.

DETAILED DESCRIPTION:
Since the introduction of Xalatan generic versions of latanoprost have entered the Canadian marketplace such as Apo-latanoprost (Apotex Inc.), Co-latanoprost (Cobalt Pharmaceuticals Co.) and Sandoz latanoprost (Sandoz Canada Inc.). The exact formulation of the different preparations of latanoprost may differ between manufacturers, although the active ingredient itself is not supposed to vary within a 15% tolerance. In a topical ocular medication in a multi-dose dispenser, the stability of the drug and its ability to penetrate the cornea into the eye may affect the efficacy of the drug.

There are no clinical trials to compare the efficacy of generic versions of latanoprost to Xalatan, nor are there any clinical trials comparing efficacy between the different generic versions. Empirical evidence based on clinical experience suggests that at least some of the generic versions of latanoprost may not be as effective as the branded version (Xalatan). Intraocular pressure is often observed to increase when switching from a branded to generic version of latanoprost, but the opposite is rarely if ever observed. The purpose of this study will be to compare the efficacy of Xalatan to two of the most popular generic versions of latanoprost available in Canada (Apo-latanoprost and Co-latanoprost).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, diagnosed with primary open angle glaucoma or ocular hypertension
* IOP currently controlled on prostaglandin analogue monotherapy (latanoprost, bimatoprost or travoprost), as judged by the investigator

Exclusion Criteria:

* Best corrected visual acuity worse than 0.6 logMAR or 20/80 Snellen in either eye.
* Patients in whom the mean IOP in either eye at the screening exam visit is greater than 36 mmHg
* History of ocular trauma within the past six (6) months.
* History of ocular infection or ocular inflammation within the past three (3) months.
* History of chronic or recurrent severe inflammatory eye disease (i.e., scleritis, uveitis)
* History of severe or serious hypersensitivity to any components of the study medications.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Intraocular surgery within the past six (6) months as determined by patient history and/or examination.
* Patients with cup/disc ratio greater than 0.80 in either eye.
* Patients with severe central visual field loss in either eye defined as a sensitivity less than or equal to 10 dB in at least two (2) of the four (4) visual field test points closest to the point of fixation. Visual field test must be within 6 months of eligibility assessment.
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Current use of ANY glucocorticoid administered by any route. Patient must have washed out of the glucocorticoid for at least 4 weeks prior to study entry.
* Use of any systemic prostaglandin or prostaglandin analogue within the last three months.
* Current use of topical non-steroidal antiinflammatory agents which inhibit cyclo-oxygenase and prostaglandin analogue synthesis.
* Any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component).
* Current use of topical non-steroidal anti inflammatory agents which inhibit cyclo-oxygenase and prostaglandin analogue synthesis.
* Angle grade less than 2 (extreme narrow angle with complete or partial closure) as measured by gonioscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 4 weeks
  Pressure within the eye will be measured at each study visit.

SECONDARY OUTCOMES:
Ocular Hyperemia | 4 weeks
  Redness of the cornea will be quantified at each study visit using the Efron scale. The scale reads 0-5, 5 being the highest level of ocular hyperemia.

CONTACTS AND LOCATIONS:
Overall Officials: David B Yan, M.D., F.R.C.S. (C), Principal Investigator — Ophthalmic Diagnostic Services
Locations (1):
- Opthalmis Diagnostic Services, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided